CLINICAL TRIAL: NCT02406690
Title: Endometrial Receptivity Profile in Patients With Endometrial Proliferation Defects
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2014-04
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Endometrial Dysfunction
Keywords: Endometrial Insufficiency; Endometrial Receptivity
MeSH Terms: interventions — Estradiol; Progesterone; Oils; Leuprolide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One tube of serum (approximately 3.5 mL) will be collected from participant at each visit via venipuncture. An uterine aspiration and endometrial biopsy sample will be taken at Day 6 of Progestrone Adminstration.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Group: Patients who failed to achieve adequate endometrial lining during a synthetic embryo transfer. This group will undergo a Leuprolide prep cycle using estradiol valerate, progesterone in oil and subsequently undergo an endometrial biopsy and uterine aspiration.
  Interventions: Other: Estradiol Valerate, Progesterone in Oil, Leuprolide
- Control Group: Patients who have achieved an adequate endometrial lining. This group will undergo a Leuprolide prep cycle using estradiol valerate, progesterone in oil and subsequently undergo an endometrial biopsy and uterine aspiration.
  Interventions: Other: Estradiol Valerate, Progesterone in Oil, Leuprolide

INTERVENTIONS:
Other: Estradiol Valerate, Progesterone in Oil, Leuprolide — Patients will undergo a Leuprolide endometrial preparatory cycle using estradiol valerate, progesterone in oil and once completed will have a uterine aspiration and biopsy performed.

SUMMARY:
The purpose of this study is to determine the differences that exist in RNA molecules, the biochemical process of methylation, and estrogen receptor binding in patients that have failed to produce adequate endometrium in synthetic embryo transfer cycles when compared to patients whose endometrium thickness is within normal limits.

DETAILED DESCRIPTION:
The purpose of this study is to determine the differences that may exist in RNA molecules, the biochemical process of methylation, and estrogen receptor binding (this is a group of proteins in the cell that are activated by the hormone estrogen) in patients that have failed to produce adequate endometrium (uterine lining) in synthetic embryo transfer cycles when compared to patients whose endometrium thickness is within normal limits.

Appropriate embryo development and luteal phase (when fertilization and implantation occur) transformation of the endometrium create a small window of opportunity where successful implantation can occur. The interaction between the embryo and the endometrium is complex and poorly understood.

The endometrium, which consists of two layers called the functionalis and basalis, goes through changes during the menstrual cycle. The changes that occur are needed for successful implantation of an embryo. The proliferative phase of the menstrual cycle is primarily governed by estrogen and is responsible for the thickening of the endometrium. Progesterone primarily controls the last half of the menstrual cycle and causes changes which allows for embryo implantation.

Through in vitro fertilization (IVF), the investigators have seen that the correct thickness of endometrium is a marker of successful implantation and ongoing pregnancy, although the reason for this is not entirely clear. In order to better understand the processes that may occur in the endometrium, the investigators are conducting a study which evaluates biochemical markers of those patients who have shown a failure to proliferate during previous synthetic IVF frozen cycles and biochemical markers of control patients who have no known endometrial pathology.

ELIGIBILITY:
Inclusion Criteria for Case Group:

* Diagnosis of endometrial insufficiency- prior cycle with maximal endometrial thickness ≤ 6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), persistent endometrial fluid.

Exclusion Criteria for Case and Control Groups:

* Any evidence for surgically induced endometrial insufficiency (Asherman's syndrome)
* Presence of hydrosalpinges that communicate with endometrial cavity
* Any contraindications to undergoing estrogen stimulation of the endometrium

  * Age ≥35 years and smoking ≥15 cigarettes per day
  * Multiple risk factors for arterial cardiovascular disease (smoking, diabetes, and hypertension)
  * Hypertension (systolic ≥140 mmHg or diastolic ≥90 mmHg)
  * Venous thromboembolism (current or history of)
  * Known thrombogenic mutations
  * Known ischemic heart disease
  * History of stroke
  * Complicated valvular heart disease (pulmonary hypertension, risk for atrial fibrillation, history of subacute bacterial endocarditis)
  * Systemic lupus erythematosus (positive or unknown antiphospholipid antibodies)
  * Migraine with aura at any age
  * Breast cancer
  * Cirrhosis
  * Hepatocellular adenoma or malignant hepatoma
  * History of undiagnosed abnormal uterine bleeding.
  * Allergic reaction to estradiol valerate, progesterone in oil, leuprolide acetate
  * Known pregnancy or delivery within the past 6 months
  * Breastfeeding
  * Obesity >35 kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who have undergone a synthetic endometrial proliferation cycle in preparation for an embryo transfer that were identified as having a proliferative phase defect will serve as the subjects. Normal, healthy patients who are undergoing infertility treatment for single gene disorder, family balancing, or male factor infertility will serve as controls. The study will occur as part of a cryosynthetic preparatory cycle prior to embryo transfer. There will be 10 cases and 10 controls recruited for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2015-09-17 (Actual); Study Completion 2015-09-17 (Actual)

PRIMARY OUTCOMES:
To determine the differences that may exist in transcriptome, methylome, and estrogen receptor binding between case and control groups | One year

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, Jr., MD, HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No